CLINICAL TRIAL: NCT01571713
Title: Patient Reported Side Effects of Pulmonary Hypertension (PH) Medications
Brief Title: Side Effects of Pulmonary Hypertension Medications
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey A. Feinstein, Principle Investigator, Stanford University
Other Study IDs: PHSE22242
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study: Pediatric patients with pulmonary hypertension

SUMMARY:
The study seeks to analyze the patient reported effects of pulmonary hypertension medications and compare these with the side effects described on the package inserts. Side effects for these PH medications have been described in the adult population, but have never been described in the pediatric population. This information can better improve patient care and be used to characterize the side effects resultant from these medications.

DETAILED DESCRIPTION:
As part of standard of care, patients are routinely asked about any symptoms they might be experiencing. This study seeks to quantify these symptoms for research purposes. Participants will be identified through those who attend the pediatric pulmonary hypertension clinic at LPCH. Only children who are currently on one of seven PH medications (Bosentan, Epoprostenol, Letairis, Sildenafil, Tadalafil, Treprostinil, Ventaris) will be approached. Patients who consent to be in the study will answer a brief series of questions pertaining to the presence and duration of their symptoms. These will be correlated to a list of side effects taken from Lexicomp (a medication database).

ELIGIBILITY:
Inclusion Criteria:

* pulmonary hypertension
* currently taking at least one of the following PH medications (Bosentan, Epoprostenol, Letairis, Sildenafil, Tadalafil, Treprostinil, Ventaris)

Exclusion Criteria:

* >18 years

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with pulmonary hypertension seen in the pulmonary hypertension clinic at Stanford Lucile Packard Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-08; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Patients Experience Side Effects | Open

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Feinstein, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No